

Joint Research Compliance Office

Centre Number (if applicable): Study Protocol Number: EudraCT number (if applicable):

## **CONSENT FORM**

Full Title of Project: Use of non-invasive optical analysis in Neurosurgery – A pilot study Date: 30/12/2019

Name of Principal Investigator: Mr Kevin O'Neill

6. I consent to take part in the above study.

| | Please initial box |
|---|---|
| 1. | I confirm that I have read and understand the participant information sheet dated 30/12/2019 version 2.0 for the above study and have had the opportunity to ask questions which have been answered fully. |
| 2. | I understand that my participation is voluntary and I am free to withdraw at any time, without giving any reason and without my medical care or legal rights being affected. |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College, from Imperial College NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. |
| 4. | I give permission for these individuals to access my records and collect clinical data that are relevant to this research. |
| 5. | I give consent for non-identifiable videos and/or images of my surgery to be collected during this study to be used in for the purpose of this research. |





Joint Research Compliance Office

| 6a. (OPTIONAL) I give consent to studies. | being contacted to potentially tak | ing part in other researc |
|---|---|---|
| Name of Patient/Participant | Signature | Date |
| Name of Person taking consent<br>(if different from Principal Investigator) | Signature | Date |
| Principal Investigator | Signature | Date |

1 copy for patient/participant; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes